CLINICAL TRIAL: NCT05189613
Title: Mepolizumab Effectiveness in Patients With Severe Eosinophilic Asthma and Co-presence of Bronchiectasis
Brief Title: Mepolizumab Effectiveness in Severe Eosinophilic Asthma and Bronchiectasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Policlinico Universitario, Catania (Other)
Responsible Party: Principal Investigator, Raffaele Campisi, Principal Investigator, Policlinico Universitario, Catania
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PoliclinicoUC
Record Dates: First submitted 2021-10-17; First posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: Bronchial Asthma; Bronchiectasis
MeSH Terms: conditions — Asthma; Bronchiectasis | interventions — mepolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Severe Asthma+BE (Experimental): Patients with severe eosinophilic asthma with co-presence of Bronchiectasis (BE) in treatment with Mepolizumab
  Interventions: Biological: Mepolizumab
- Severe Asthma without BE (Active Comparator): Patients with severe eosinophilic asthma without Bronchiectasis (BE) in treatment with Mepolizumab
  Interventions: Biological: Mepolizumab

INTERVENTIONS:
Biological: Mepolizumab — Subcutaneous Mepolizumab (100 mcg) injection in patients with severe eosinophilic asthma

SUMMARY:
Asthma is a chronic respiratory disorder characterized by bronchial inflammation and reversible bronchial obstruction. Severe asthma is an extremely heterogeneous disease, often associated with several comorbidities and risk factors. Severe uncontrolled asthma associated with bronchiectasis is an emerging phenotype. Several studies have attempted to establish an association between asthma and bronchiectasis. Mepolizumab, an Interleukin-5 (IL-5) antagonist, reduces exacerbations, eosinophils, and improves pulmonary function and asthma control. IL-5 is pivotal to eosinophils maturation and release from bone marrow, their subsequent accumulation, activation and persistence in the tissues. IL-5 therefore represents an attractive target to prevent or blunt eosinophils-mediated inflammation. The investigators hypothesize that eosinophils, stimulated by IL-5, play a crucial role in severe asthma and BE pathogenesis.

DETAILED DESCRIPTION:
Asthma is a chronic respiratory disorder in which bronchial inflammation, airway hyperresponsiveness, and reversible bronchial obstruction are operant, inciting daily symptoms and triggering unpredictable acute exacerbations. The prevalence of severe asthma varies between 5 and 10% of asthma frameworks and is estimated to account for >60% of the total costs of the disease. Severe asthma warrants Global Initiative for Asthma (GINA) Step 4 or 5 treatment, (e.g. high-dose Inhaled Corticosteroids/Long Acting Beta2-Agonists (ICS/LABA), to achieve control or remains 'uncontrolled' (entirely or in part) despite this or other appropriate therapeutic intervention. Severe asthma is an extremely heterogeneous disease, often associated with several comorbidities and risk factors, leading to divide accordingly severe asthmatic patients into homogenous groups. The result is the identification of several phenotypes of severe asthma, as those associated with obesity, smoking habit, chronic obstructive pulmonary disease (COPD), gastro-oesophageal reflux disease (GERD), chronic rhinosinusitis, nasal polyposis, infections and others. In recent years, the recognition and treatment of comorbidities is crucial because can potentially improve asthma control and outcomes. Severe uncontrolled asthma associated with bronchiectasis is an emerging phenotype. Several studies have attempted to establish an association between asthma and bronchiectasis. The prevalence of bronchiectasis (BE) is significantly higher in severe asthma (range 24-40%), then in milder disease (3%). At least one third of patients with severe asthma show the presence of BE on high resolution chest computed tomography (HRCT) scan. This phenotype has been described particularly in patients with severe, late-onset eosinophilic asthma. In order to improve the therapeutic approach to the more severe forms of asthma, biological treatments have been realized. Recently, mepolizumab, an IL-5 antagonist, was commercialized. Mepolizumab reduces exacerbations, eosinophils, and improves pulmonary function and asthma control. There is a considerable evidence that implicates eosinophils as important effector cells in the eosinophilic asthma inflammation. IL-5 is pivotal to eosinophils maturation and release from bone marrow, their subsequent accumulation, activation and persistence in the tissues. IL-5 therefore represents an attractive target to prevent or blunt eosinophils-mediated inflammation. The investigators hypothesize that eosinophils, stimulated by IL-5, play a crucial role in severe asthma and BE pathogenesis. Accumulation of eosinophils at the bronchial level causes damage by degranulation and release of toxic protein, mucus hypersecretion, elastolytic activity, mucinous cells hypertrophy and oxidative stress. Airway remodeling, due to the activity of eosinophils, is the consequence of ongoing inflammation and repair. All these tissue changes are characteristic of both asthma and bronchiectasis (BE). BE, in effect, is caused by long-term excessive inflammatory damage to the airways and in patients with asthma, eosinophils may further contribute to tissue injury. The investigators therefore hypothesize that treatment with mepolizumab, targeted against IL-5 activity, in patients with severe eosinophilic asthma associated with bronchiectasis may lead to a reduction of bronchiectasis and asthma exacerbations and lead to improve control of asthma.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female with age greater than or equal to 18 years;
2. Severe eosinophilic asthma diagnosis according to GINA 2019 report
3. Evidence of bronchiectasis in at least one lung lobe in the chest CT scan performed prior to mepolizumab treatment;
4. Presence of daily expectoration;
5. At least 3 bronchiectasis exacerbations in the year prior to mepolizumab treatment, documented through medical documentation, which required treatment with antibiotics;
6. Informed consent obtained from the patient.

Exclusion Criteria:

1. Poor adherence to severe asthma therapy
2. Patients with other respiratory disease that may share common clinical manifestations of severe asthma (i.e. acute bronchopulmonary aspergillosis, vasculitis and COPD)
3. Any medical condition or disease that was not stable during the 3 months prior to mepolizumab treatment (excluding asthma exacerbations), that the investigator believes may compromise the safety of the patient if enrolled in the study such us atrial fibrillation, acute respiratory failure, acute heart failure, myocardial infarction and acute renal failure.
4. Bronchiectasis associated with cystic fibrosis;
5. Traction bronchiectasis in the context of pulmonary fibrosis;
6. History of lung cancer in the previous 5 years;
7. History of significant hemoptysis (≥300 mL of blood) or which required embolization or blood transfusions within 6 weeks prior to mepolizumab treatment;
8. Use of drugs that can influence the response to treatment such us immunosuppressant and/or biological therapies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of Asthma Control Test (ACT) score at Week 12 (T3), at Week 24 (T6) and at Week 52 (T12). | Baseline and Week 52
  Asthma Control Test (ACT) score is validated five-points scoring system, self-administered assessing the control of Asthma.
  Scores range from 5 points (worst asthma control) to 25 points (better asthma control).
  Change = Week 12 (T3) - Baseline score; Week 24 (T6) - Baseline score; Week 52 (T12) - Baseline score.

SECONDARY OUTCOMES:
Change from Baseline values of Spirometry values (expressed in Litre) at Week 12 (T3), at Week 24 (T6) and at Week 52 (T12). | Baseline and Week 52
  Spirometry assess the airways obstruction. Spirometry will be performed according to American Thoracic Society (ATS)/European Respiratory Society (ERS) guidelines.
  The main benchmarks for assessing airways obstruction are: Forced Expiratory Volume in 1 second (FEV1) and Forced Vital Capacity (FVC), expressed in Litre (L) respectively.
  Change = Week 12 (T3) - Baseline values; Week 24 (T6) - Baseline values; Week 52 (T12) - Baseline values.

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele Campisi, Medicine, Principal Investigator — Respiratory Unit Policlinico G. Rodolico-San Marco
Locations (1):
- AOU Policlinico "G. Rodolico-Sto arrivando!n Marco", Catania, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chung KF, Wenzel SE, Brozek JL, Bush A, Castro M, Sterk PJ, Adcock IM, Bateman ED, Bel EH, Bleecker ER, Boulet LP, Brightling C, Chanez P, Dahlen SE, Djukanovic R, Frey U, Gaga M, Gibson P, Hamid Q, Jajour NN, Mauad T, Sorkness RL, Teague WG. International ERS/ATS guidelines on definition, evaluation and treatment of severe asthma. Eur Respir J. 2014 Feb;43(2):343-73. doi: 10.1183/09031936.00202013. Epub 2013 Dec 12. PMID 24337046
- [Result] Crimi C, Campisi R, Cacopardo G, Intravaia R, Nolasco S, Porto M, Pelaia C, Crimi N. Real-life effectiveness of mepolizumab in patients with severe refractory eosinophilic asthma and multiple comorbidities. World Allergy Organ J. 2020 Sep 18;13(9):100462. doi: 10.1016/j.waojou.2020.100462. eCollection 2020 Sep. PMID 32994855
- [Result] Bardin PG, Rangaswamy J, Yo SW. Managing comorbid conditions in severe asthma. Med J Aust. 2018 Jul 16;209(S2):S11-S17. doi: 10.5694/mja18.00196. PMID 30453867
- [Result] Perez-Miranda J, Traversi L, Polverino E. Bronchiectasis in severe asthma: a distinct phenotype? Curr Opin Pulm Med. 2019 Jan;25(1):71-78. doi: 10.1097/MCP.0000000000000542. PMID 30461531
- [Result] Carpagnano GE, Scioscia G, Lacedonia D, Curradi G, Foschino Barbaro MP. Severe uncontrolled asthma with bronchiectasis: a pilot study of an emerging phenotype that responds to mepolizumab. J Asthma Allergy. 2019 Mar 5;12:83-90. doi: 10.2147/JAA.S196200. eCollection 2019. PMID 30881051
- [Result] Padilla-Galo A, Olveira C, Fernandez de Rota-Garcia L, Marco-Galve I, Plata AJ, Alvarez A, Rivas-Ruiz F, Carmona-Olveira A, Cebrian-Gallardo JJ, Martinez-Garcia MA. Factors associated with bronchiectasis in patients with uncontrolled asthma; the NOPES score: a study in 398 patients. Respir Res. 2018 Mar 16;19(1):43. doi: 10.1186/s12931-018-0746-7. PMID 29548297
- [Result] Dimakou K, Gousiou A, Toumbis M, Kaponi M, Chrysikos S, Thanos L, Triantafillidou C. Investigation of bronchiectasis in severe uncontrolled asthma. Clin Respir J. 2018 Mar;12(3):1212-1218. doi: 10.1111/crj.12653. Epub 2017 Jun 8. PMID 28544140
- [Result] Pelaia C, Crimi C, Vatrella A, Tinello C, Terracciano R, Pelaia G. Molecular Targets for Biological Therapies of Severe Asthma. Front Immunol. 2020 Nov 30;11:603312. doi: 10.3389/fimmu.2020.603312. eCollection 2020. PMID 33329598
- [Result] Pelaia C, Crimi C, Pelaia G, Nolasco S, Campisi R, Heffler E, Valenti G, Crimi N. Real-life evaluation of mepolizumab efficacy in patients with severe eosinophilic asthma, according to atopic trait and allergic phenotype. Clin Exp Allergy. 2020 Jul;50(7):780-788. doi: 10.1111/cea.13613. Epub 2020 May 13. PMID 32347992
- [Result] Polverino E, Dimakou K, Hurst J, Martinez-Garcia MA, Miravitlles M, Paggiaro P, Shteinberg M, Aliberti S, Chalmers JD. The overlap between bronchiectasis and chronic airway diseases: state of the art and future directions. Eur Respir J. 2018 Sep 15;52(3):1800328. doi: 10.1183/13993003.00328-2018. Print 2018 Sep. PMID 30049739
- [Result] Kaur R, Chupp G. Phenotypes and endotypes of adult asthma: Moving toward precision medicine. J Allergy Clin Immunol. 2019 Jul;144(1):1-12. doi: 10.1016/j.jaci.2019.05.031. PMID 31277742